CLINICAL TRIAL: NCT01774292
Title: Evaluation of the Effect of Intracuff Alkalinized Lidocaine on Coughing Incidence at Extubation in Surgeries Without Nitrous Oxide Lasting More Than 2 Hours
Brief Title: Effect of Intracuff Alkalinized Lidocaine on Coughing Incidence at Extubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Yanick Sansoucy, Anesthesiologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12182
Record Dates: First submitted 2013-01-04; First posted 2013-01-23 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Coughing; Extubation; Lidocaine; Endotracheal Cuff
Keywords: Impact of alkalized lidocaine on coughing at extubation
MeSH Terms: conditions — Cough | interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alkalized lidocaine (Active Comparator): 160 mg of 4% lidocaine (4 ml) in the endotracheal cuff and add bicarbonate 8,4% until appropriate seal.
  Interventions: Procedure: Endotracheal intubation with injection of liquid in the cuff
- Sterile saline (Placebo Comparator): 4 mL of sterile saline in the endotracheal cuff and add bicarbonate 8,4% until appropriate seal.
  Interventions: Procedure: Endotracheal intubation with injection of liquid in the cuff

INTERVENTIONS:
Procedure: Endotracheal intubation with injection of liquid in the cuff

SUMMARY:
The purpose of the study is to determined whether the administration of alkalized 4% lidocaine (160 mg) in the endotracheal tube cuff is effective in diminishing the incidence of coughing at extubation in surgeries lasting more than 2 hours without the use of nitrous oxide as an anesthetic agent.

DETAILED DESCRIPTION:
The diffusion of nitrous oxide inside the endotracheal cuff leads to increase pressure, pain and coughing. Studies have shown benefit of alkalized lidocaine and other mediums within the cuff with nitrous oxide. No study has yet evaluated the benefit of alkalized lidocaine in long surgeries without the use of nitrous oxide.

ELIGIBILITY:
Inclusion Criteria:

- ASA 1,2 or 3 patients requiring general anesthesia for an elective urological or gynecological surgery predicted to last more than 2 hours

Exclusion Criteria:

* Patient refusal
* Lidocaine allergy
* Any allergies to drugs or anesthetics used during the study
* Under 18 years of age
* Pregnant
* Previous airway surgery
* Cormack 3 or 4 or anticipated difficult airway
* Upper respiratory tract infection in the last month
* Active respiratory disease
* Chronic cough or throat pain
* Gastro-esophageal reflux disease or at risk for aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Coughing | 24 hours after the end ofsurgery

SECONDARY OUTCOMES:
Throat pain | 24 hours after the end of surgery
Nausea and Vomiting | 24 hours after end of surgery
Hoarseness of the voice | 24 hours after end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanick Sansoucy, Doctor, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Estebe JP, Delahaye S, Le Corre P, Dollo G, Le Naoures A, Chevanne F, Ecoffey C. Alkalinization of intra-cuff lidocaine and use of gel lubrication protect against tracheal tube-induced emergence phenomena. Br J Anaesth. 2004 Mar;92(3):361-6. doi: 10.1093/bja/aeh078. PMID 14970135
- [Background] Estebe JP, Gentili M, Le Corre P, Dollo G, Chevanne F, Ecoffey C. Alkalinization of intracuff lidocaine: efficacy and safety. Anesth Analg. 2005 Nov;101(5):1536-1541. doi: 10.1213/01.ANE.0000180995.24211.89. PMID 16244028
- [Background] Estebe JP, Dollo G, Le Corre P, Le Naoures A, Chevanne F, Le Verge R, Ecoffey C. Alkalinization of intracuff lidocaine improves endotracheal tube-induced emergence phenomena. Anesth Analg. 2002 Jan;94(1):227-30, table of contents. doi: 10.1097/00000539-200201000-00044. PMID 11772834
- [Background] Dollo G, Estebe JP, Le Corre P, Chevanne F, Ecoffey C, Le Verge R. Endotracheal tube cuffs filled with lidocaine as a drug delivery system: in vitro and in vivo investigations. Eur J Pharm Sci. 2001 Jun;13(3):319-23. doi: 10.1016/s0928-0987(01)00119-1. PMID 11384855
- [Background] Navarro LH, Lima RM, Aguiar AS, Braz JR, Carness JM, Modolo NS. The effect of intracuff alkalinized 2% lidocaine on emergence coughing, sore throat, and hoarseness in smokers. Rev Assoc Med Bras (1992). 2012 Mar-Apr;58(2):248-53. PMID 22569622
- [Derived] Souissi H, Frechette Y, Murza A, Masse MH, Marsault E, Sarret P, D'Aragon F, Parent AJ, Sansoucy Y. Intracuff 160 mg alkalinized lidocaine reduces cough upon emergence from N2O-free general anesthesia: a randomized controlled trial. Can J Anaesth. 2016 Jul;63(7):862-70. doi: 10.1007/s12630-016-0652-8. Epub 2016 Apr 13. PMID 27075030